CLINICAL TRIAL: NCT07301567
Title: A Proof-of-concept Pilot Study to Determine the Safety and Effectiveness of the Negative Pressure Neck Therapy (NPNT) in Healthy Participants.
Brief Title: Pilot Study of Negative Pressure Neck Therapy (NPNT)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other)
Responsible Party: Principal Investigator, John Fleetham, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: H25-02563
Record Dates: First submitted 2025-11-25; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Apnea; Sleep Apnea Syndrome, Obstructive; Sleep Disorder (Disorder)
Keywords: sleep apnea; Obstructive sleep apnea; sleep disordered breathing
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Wake Disorders; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): One night of Home sleep apnea testing (HSAT) with Negative Pressure Neck Therapy (NPNT) intervention, followed by 7 night washout, then one night of HSAT only
  Interventions: Device: Negative Pressure Neck Therapy (NPNT)
- Group 2 (Experimental): One night of HSAT only, followed by 7 night washout, then one night of HSAT with NPNT intervention.
  Interventions: Device: Negative Pressure Neck Therapy (NPNT)

INTERVENTIONS:
Device: Negative Pressure Neck Therapy (NPNT) — Negative pressure neck therapy (NPNT) is a self-contained, non-invasive, soft, flexible, external neck collar

SUMMARY:
Obstructive sleep apnea (OSA) is a serious, chronic sleep-related breathing disease in which the upper airway repeatedly collapses during sleep, leading to intermittent oxygen deprivation. This pilot study will evaluate the Safety and Efficacy of Negative Pressure Neck Therapy (NPNT) in up to 10 healthy participants. Participants will undergo 2 separate home sleep apnea tests (HSAT) approximately 1 week apart and will be randomly assigned to wear the NPNT device at either night 1 or night 2 of HSAT. Participation will include 5 on-site visits and 1 phone call over approximately 1 month.

DETAILED DESCRIPTION:
Purpose: To determine the safety and efficacy of the Negative Pressure Neck Therapy (NPNT) in Healthy Participants.

Negative pressure neck therapy (NPNT) uses a self-contained, non-invasive, external device to apply a gentle, outward pulling effect around the neck's surface.

Hypothesis: Given the exploratory nature and small sample size no formal hypothesis testing will be conducted

Objectives:

Primary Objective:

1. To determine if NPNT can effectively reduce the number of apnea-hypopnea index (AHI) events (sleep disorder breathing events) in healthy participants.

Secondary Objectives:

1. To determine the tolerability of the NPNT
2. To determine the duration of time required for acclimating to the device
3. To determine the NPNT parameters (optimal device fit) based on participant characteristics.
4. To collect feedback from participants regarding the device use, comfort, fit, function, usability, etc.

Safety and Efficacy Objectives:

1. To evaluate the safety and effectiveness of NPNT
2. To assess potential side effects of NPNT.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≤42 kg/m2
* Able to speak, read, and write English

Exclusion Criteria:

* Known sleep disorder such as Obstructive Sleep Apnea (OSA), narcolepsy, restless leg syndrome, idiopathic hypersomnolence or chronic insomnia
* No previous surgery, injury, or radiation to the neck
* Excessive hair or beard in the area of the neck, and/or unwillingness to shave that area for the duration of this study
* Inflammatory skin condition, such as acne or eczema in the neck area
* Known silicone allergy
* Night shift work because of irregular sleep-wake cycles
* Excessive alcohol intake, defined as that leading to interference with work, home life, or the ability to optimally perform normal everyday duties and tasks
* Use of illicit drugs currently or within the past 5 years
* Serious pulmonary disease
* Use of home oxygen or oxygen saturation <94%
* Cancer that has been in remission for less than one year
* Previous surgery for peripheral arterial disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of the number of sleep-disordered breathing events between intervention and control nights as assessed by Home Sleep Apnea Test (HSAT). | 1 night
  Change between control night and intervention night on mean AHI (Apnea-Hypopnea Index) scores. A positive treatment effect will be attributed to the NPNT device if the difference between the mean AHI score on intervention night is less than the mean AHI score on control night. A score of less than 0 is positive.
  Measurement Tool: HSAT (Home Sleep Apnea Test) Unit of Measure: AHI (Apnea-Hypopnea Index) scores

SECONDARY OUTCOMES:
Tolerability of NPNT device based on duration of time (hours) worn during NPNT intervention night as assessed by Participant Report and Home Sleep Apnea Test (HSAT) | 1 night
  Wear time (hours) of NPNT device will be assessed for each participant during the NPNT intervention night, after 7 day NPNT acclimatization period. Mean, median, range of tolerability of scores will be reported.
  Measurement Tool: Participant Reported and HSAT (Home Sleep Apnea Test) Unit of Measure: hours
Participant Characteristics will be assessed compared to NPNT device fit/shape based on participant response on the Device Evaluation Questionnaire using Likert scores. | 1 night
  Descriptive participant traits (age, BMI, craniofacial markers, etc.) will plotted against NPNT device fit/shape Likert scores from the Device Evaluation Questionnaire above and below a score of 3. For example, fit/shape Likert score rating by BMI category.
  Measurement Tool: Device Evaluation Questionnaire and Participant demographics Unit of Measure: Likert Score
Participant reported device tolerability will be assessed using the Device Evaluation Questionnaire Likert scale responses. | 1 night
  Proportion of participants rating NPNT device as "tolerable" (≥3 on Likert scale) during NPNT intervention night, after 7 day acclimatization period.
  Measurement Tool: Device Evaluation Questionnaire Unit of Measure: Likert scale
Participant Reported Feedback on shape and fit of NPNT device as assessed by the Device Evaluation Questionnaire using a Likert Scale (≥3 on Likert scale) | 1 night
  Proportion of participants rating device as "Moderate/good/excellent" (e.g., ≥3 on Likert scale). Mean, median, range of shape/fit scores, including a breakdown by demographic/ BMI group will be assessed after NPNT intervention night and 7 day acclimatation period.
  Measurement Tool: Device Evaluation Questionnaire Unit of Measure: Likert scale
Participant Feedback on NPNT device comfort, usability and function based on the Device Evaluation Questionnaire using a Likert scale | 1 night
  Proportion of participants rating device comfort, usability and function as ≥3 on Likert scale. Mean, median, range of device comfort, usability and function scores, including a breakdown by demographic/ BMI group will be assessed after NPNT intervention night and after 7 day acclimatation period.
  Measurement Tool: Device Evaluation Questionnaire Unit of Measure: Likert scale
Participant Feedback on NPNT device based on qualitative data (open comments) from the Device Evaluation Questionnaire after the NPNT device intervention night. | 1 night
  Qualitative data will be summarized using simple thematic coding based on participant open comment section of the Device Evaluation Questionnaire after the NPNT device intervention night, after 7 day acclimatization period.
  Measurement Tool: Device Evaluation Questionnaire Unit of Measure: Qualitative data (open comments)

OTHER OUTCOMES:
Adverse Events based on Device Evaluation Questionnaire responses to adverse device effects after NPNT intervention night and 7 night acclimatization period. | 8 nights
  Device specific adverse events (skin irritation, redness or rash, discomfort or pain, swelling, other) will be assessed using a scale of 1 to 5 (not at all, mild, moderate, severe, very severe) after the NPNT intervention night and 7 night acclimatization period.
  Measurement Tool: Device Evaluation Questionnaire Unit of Measure: Scale of 1-5 (1-not at all, 2-mild, 3-moderate, 4-severe, 5-very severe)

CONTACTS AND LOCATIONS:
Overall Officials: John A Fleetham, MD, Principal Investigator — VCHA/UBC
Locations (2):
- Canada (2):
  - Centre for Lung Health, Vancouver, British Columbia
  - Leon Judah Blackmore Centre for Sleep Disorders, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Undecided
This is a pilot study, so only IPD used in the results publication may be shared in the future.